CLINICAL TRIAL: NCT03279939
Title: Evaluation of Heidelberg Engineering SPECTRALIS With OCT Angiography Module
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: S-2017-1
Record Dates: First submitted 2017-09-04; First posted 2017-09-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Retinal Vascular; Normal Eyes
MeSH Terms: interventions — Fluorescein Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Subjects with Normal Eyes: OCT Angiography, Color Fundus Photography, and Fluorescein Angiography as per protocol in subjects without ophthalmic pathology.
  Interventions: Device: OCT Angiography; Device: Color Fundus Photography; Device: Fluorescein Angiography
- Subjects with Pathology: OCT Angiography, Color Fundus Photography, Fluorescein Angiography, and when clinically indicated, Indocyaine Green Angiography as per protocol in subjects with retinal vascular pathology.
  Interventions: Device: OCT Angiography; Device: Color Fundus Photography; Device: Fluorescein Angiography; Device: Indocyaine Green Angiography

INTERVENTIONS:
Device: OCT Angiography — OCT Angiography offers clinicians a non-invasive three-dimensional visualization of vasculature in the retina and choroid. The visualization of perfused vasculature in a three-dimensional layout, offers clinicians an aid in the identification of retinal and choroidal pathologies such as retinal ischemia, microaneurysms, retinal neovascularization and choroidal neovascular membranes.
  Other Names: OCTA
Device: Color Fundus Photography — Non-contact white light photography.
  Other Names: CFP
Device: Fluorescein Angiography — An imaging procedure where dye is injected into a vein and images are taken of the back of the eye to visualize the perfusion of retinal vessels in two dimensional images.
  Other Names: FA
Device: Indocyaine Green Angiography — An imaging procedure where dye is injected into a vein and images are taken of the back of the eye to visualize the perfusion of choroidal vessels in two dimensional images.
  Other Names: ICGA
  Groups: Subjects with Pathology

SUMMARY:
Assessment of image quality and clinical relevance of OCT Angiography via comparison to FA/ICGA.

DETAILED DESCRIPTION:
The objectives of this study are:

1. To compare the OCTA image quality between the SPECTRALIS and the predicate.
2. To compare the agreement of clinical findings on SPECTRALIS OCTA to the predicate.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Able and willing to undergo the test procedures, sign informed consent, and follow instructions.
* Age ≥ 22

Subjects with Normal Eyes:

* Subjects presenting at the site without uncontrolled systemic conditions, or ocular disease, as determined by the Investigator
* Corrected visual acuity ≥ 20/40 in each eye
* No history of ocular surgical intervention (except for refractive or cataract surgery) in either eye

Subjects with Pathology:

* Subjects with retinal conditions in at least one eye.
* Subjects included can have a range of retinal vascular pathologies affecting different anatomic depths through the retina and choroid. Retinal conditions including but not limited to diabetic retinopathy, wet age-related macular degeneration (AMD), and branch or central retinal vein occlusion that give rise to features such as retinal ischemia, microaneurysms, choroidal neovascularization and retinal neovascularization will be included.

Exclusion Criteria:

* Subjects unable to read or write
* Subjects with ocular media not sufficiently clear to obtain acceptable study-related imaging
* Subjects who cannot tolerate the imaging procedures
* Subjects with known allergies to fluorescein dye, Indocyanine Green (ICG), shellfish, drugs for pupillary dilation
* Subjects with contraindication to pupillary dilation in study eye

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with Normal Eyes:
  * Subjects presenting at the site without uncontrolled systemic conditions, or ocular disease, as determined by the Investigator
  * Corrected visual acuity ≥ 20/40 in each eye
  * No history of ocular surgical intervention (except for refractive or cataract surgery) in either eye
  Subjects with Pathology:
  * Subjects with retinal conditions in at least one eye.
  * Subjects included can have a range of retinal vascular pathologies affecting different anatomic depths through the retina and choroid. Retinal conditions including but not limited to diabetic retinopathy, wet age-related macular degeneration (AMD), and branch or central retinal vein occlusion that give rise to features such as retinal ischemia, microaneurysms, choroidal neovascularization and retinal neovascularization will be included.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
OCTA image quality | day 1
  Image quality grading results of study selected images
Clinically relevant findings on OCTA | day 1
  Clinically relevant grading results of study selected images

CONTACTS AND LOCATIONS:
Overall Officials: David Brown, MD, Principal Investigator — Retina Consultants Houston
Locations (1):
- Retina Consultants of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No